CLINICAL TRIAL: NCT03867890
Title: Is Consumer Behaviour Towards Footwear Predisposing for Lower Extremity Injuries in Runners and Walkers? A Prospective Study
Brief Title: Relationship Between Footwear Consumer Behaviour and Lower Extremity Injuries
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201214347
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Risk Factor; Sports Injury; Footwear
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
A prospective cohort study was set-up in leisure-time walkers and runners. Potential risk factors in consumer behaviour were obtained by means of a baseline questionnaire related to the acquisition of current walking or running shoes. Information on injuries sustained during a 24 week period after the baseline questionnaire was obtained in 104 runners and 104 walkers using a 2-weekly questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* walk or run at least 10 kilometres per week
* maintain a minimal distance of ten kilometres per week, for a period of 24 weeks
* wear one and the same pair of shoes during walking/running activities during this period

Exclusion Criteria:

* systemic disease, cardiac problems or diabetes
* complaints at the lower extremities in the last two weeks,
* surgery at the lower extremities in the last three years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Leisure-time runners and walkers
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
injury occurence | 24 weeks
  self-reported running or walking injury questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep Revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided